CLINICAL TRIAL: NCT02310659
Title: Study to Evaluate the Association of Testosterone Levels With Coronary Artery in Patients With Stable Coronary Artery Disease
Brief Title: Study to Evaluate the Association of Testosterone Levels With Coronary Artery Calcification
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Jiangtao Lai, MD, Zhejiang University
Other Study IDs: 20090206
Record Dates: First submitted 2014-12-01; First posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- lower calcificant score group: patients with coronary artery calcificant score <400
  Interventions: Other: No intervention
- higher calcificant score group: patients with coronary artery calcificant score ≥400
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Coronary artery calcification (CAC) is a pandemic condition in elderly patients with coronary artery disease (CAD) and associated with worse prognosis. Although available data shows association between testosterone levels in men and CAD, the association between testosterone and CAC in old-aged male patients with CAD remains unknown. In this study, the relationship of serum testosterone levels with CAC score in elderly male patients with CAD was evaluated.

DETAILED DESCRIPTION:
Coronary artery calcification (CAC) is associated with worse outcomes in patients with coronary artery disease (CAD), especially in old-aged population. Extensive CAC also increases the risk of procedure associated complications, such as stent migration, coronary artery perforation, dissection and thrombosis. The pathogenesis of CAC has not been fully explained. Recent evidence suggests that CAC share common pathways with bone formation. So, it can be presumed that risk factors contributing to bone formation and resorption activity also affect the development of CAC. Sex hormones is known to play an important role in bone development and in bone quality maintenance. Available data shows that androgens may affect differentiation, proliferation, and apoptosis of osteocytes, osteoclasts, and osteoblasts. Androgen receptor expression has been detected on different types of cells which contributing to the bone formation, such as osteoblastes, osteocytes and condrocytes, and androgen deprivation therapy results negative effects on bone mineral density in patients with metastatic prostate cancer. Osteoporosis, a systemic disease characterized by bone tissue loss, is more prevalent in oler men with low testosterone levels. In CAC, pathophysiological researches show that several vascular cell types, such as vascular smooth muscle cells, adventitial myofibroblasts and microvascular pericytes, have the potential to produce mineralized matrix and differentiate into osteoblasts. So, it can be postulated that androgens may play a similar role in the development of CAC.

Up to date, only limited data is available about the association between testosterone and CAC. A single-center study with relatively small sample revealed an inverse association between testosterone and CAC in non-obese men. The aim of this study was to investigate the association between testosterone and CAC measured as CAC score in old-aged male patients with CAD.

ELIGIBILITY:
Inclusion Criteria:

* Elderly male patients (age ≥ 65 years old) with stable angina and proven coronary artery disease

Exclusion Criteria:

* Less than 65 years old
* Acute coronary syndrome
* History of PCI or coronary artery bypass grafting
* History of myocardial infarction
* Renal dysfunction defined by glomerular filtration rate < 30 mL/min

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly male patients (age ≥ 65 years old) with stable angina and proven coronary artery disease
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with severe coronary artery calcification | 10 months
  Number of participants with coronary artery calcification score ≥400

CONTACTS AND LOCATIONS:
Overall Officials: Junzhu Chen, MD, Study Chair — Zhejiang University
Locations (1):
- 1st Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China